CLINICAL TRIAL: NCT01996059
Title: A Multi-center Pilot Randomized Controlled Trial Examining the Differences of Nutritional Status of Patients Undergoing Functional Jejunal Interposition Or Roux-en-Y After Total Gastrectomy for Gastric Cancer
Brief Title: Functional Jejunal Interposition Improve Nutritional Status After Total Gastrectomy
Acronym: FJINS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Junsheng Peng,MD, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012017
Record Dates: First submitted 2013-11-19; First posted 2013-11-27 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Gastric Cancer; Nutrition Disorders
Keywords: nutritional status; functional jejunal interposition; Roux-en-Y; gastrectomy
MeSH Terms: conditions — Stomach Neoplasms; Nutrition Disorders | interventions — Anastomosis, Roux-en-Y

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Functional Jejunal Interposition (Experimental): First, an end-to-side esophagojejunostomy was performed at 40 cm anal to Treitz's ligament. Then, an end-to-side duodenojejunostomy was created at the efferent limb 35 cm distal to the esophagojejunostomy, followed by a side-to-side jejunostomy at 5 cm distal to duodenojejunostomy and 20 cm distal to Treitz's ligament. Finally, 2 jejunal proper ligations were made at 5 cm oral to esophagojejunostomy and 2 cm distal to duodenojejunostomy.
  Interventions: Procedure: Functional Jejunal Interposition
- Roux-en-Y (Active Comparator): The distal end of the duodenum was closed. The jejunum was separated 15-20cm distal to the Treitz's ligament, and an end-to-side esophagojejunostomy was done at the distal side of the jejunum. Then, the continuity of the jejunum was reconstructed with side-to-end jejunojejunostomy at 40-45cm distal to esophagojejunostomy.
  Interventions: Procedure: Roux-en-Y

INTERVENTIONS:
Procedure: Functional Jejunal Interposition — First, an end-to-side esophagojejunostomy was performed at 40 cm anal to Treitz's ligament. Then, an end-to-side duodenojejunostomy was created at the efferent limb 35 cm distal to the esophagojejunostomy, followed by a side-to-side jejunostomy at 5 cm distal to duodenojejunostomy and 20 cm distal to Treitz's ligament. Finally, 2 jejunal proper ligations were made at 5 cm oral to esophagojejunostomy and 2 cm distal to duodenojejunostomy.
  Arms: Functional Jejunal Interposition
Procedure: Roux-en-Y — The distal end of the duodenum was closed. The jejunum was separated 15-20cm distal to the Treitz's ligament, and an end-to-side esophagojejunostomy was done at the distal side of the jejunum. Then, the continuity of the jejunum was reconstructed with side-to-end jejunojejunostomy at 40-45cm distal to esophagojejunostomy.
  Arms: Roux-en-Y

SUMMARY:
The purpose of this study is to find out whether the nutritional status of patients undergoing Functional Jejunal Interposition is better than those with Roux-en-Y After Total Gastrectomy for Gastric Cancer. To find a better reconstruction for patients who received total gastrectomy.

DETAILED DESCRIPTION:
Surgery is the only curative way for gastric cancer to date. Methods of Resection and reconstruction are closely related to prognosis and nutritional status. Therefore, it is essential to choose. At present, more and more clinical centers tend to choose Roux-en-Y (RY) reconstruction after total gastrectomy, which are prone to a variety of complications, and seriously affects the quality of life, such as malnutrition. There is argument over whether functional jejunal interposition is better than those with Roux-en-Y After total gastrectomy for gastric cancer. How to improve the nutritional status of the patients following total gastrectomy with gastrointestinal reconstruction arouses people's attention. The purpose of this study was to evaluate differences of the nutritional status in patients undergoing functional jejunal interposition and Roux-en-Y after total gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Untreated patients with curative resectable gastric cancer (A)a clear pathological diagnosis (B)the surgeon and radiologist assess the possibility of removal (C)no previous history of other malignancies. (D)the patient has signed an informed consent form (E)cardiopulmonary and kidney function is normal (F)ECOG body condition scores 0 to 1 (G)does not require emergency surgery

Exclusion Criteria:

- (A) pregnant or lactating women; (B) of the liver, lung, bone, and other distant metastasis; (C) positive supraclavicular lymph nodes, pelvic or ovarian species, peritoneal dissemination, etc.; (D) massive ascites, cachexia; (E) with other serious diseases, including cardiovascular, respiratory, kidney, or liver disease, poor merger control hypertension, diabetes; (F) mental disorder or disease; (G) 4 weeks prior to enrollment participated or are participating in other clinical trials of patients; (H) had undergone surgery, and its influence has not been eliminated for patients; (I) a history of stomach or esophagus cancer, including stromal tumors, sarcoma, lymphoma, carcinoid; (J) combined with active infection in patients (infection caused by fever above 38 ℃); (K) in patients with poor compliance or poor patient compliance investigators to consider; (L) Some researchers believe that other clinical, laboratory conditions patients should not participate in the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2012-07; Primary Completion 2020-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index | 3 months

SECONDARY OUTCOMES:
Onodera Prognosis Nutritional Index | 3 months

OTHER OUTCOMES:
Visick rates | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Junsheng Peng, professor, Principal Investigator — Department of Gastrointestinal Surgery
Locations (1):
- the 6th Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China